CLINICAL TRIAL: NCT00444925
Title: 12-Week, Randomized, Double-Blind, Double-Dummy,Placebo-Controlled, Parallel-Group, Multicenter Trial To Evaluate The Efficacy And Safety Of Fesoterodine In Comparison To Tolterodine ER In Patients With Overactive Bladder (OAB)
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Fesoterodine in Comparison to Tolterodine for Overactive Bladder (OAB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221008
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fesoterodine (Experimental): Tablets
  Interventions: Drug: fesoterodine fumarate
- Placebo (Placebo Comparator): Tablets and capsules
  Interventions: Drug: placebo
- Tolterodine (Active Comparator): Capsules
  Interventions: Drug: tolterodine tartrate

INTERVENTIONS:
Drug: fesoterodine fumarate — 4 mg once daily (OD) for 1 week followed by a forced dose-escalation to 8 mg once daily (OD) for 11 weeks
  Arms: Fesoterodine
Drug: placebo — once daily (OD)for 12 weeks
  Arms: Placebo
Drug: tolterodine tartrate — 4 mg once daily (OD) for 12 weeks
  Arms: Tolterodine

SUMMARY:
To evaluate the efficacy and safety of fesoterodine in comparison to tolterodine and placebo for overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Adult overactive bladder (OAB) patients who present with OAB symptoms, including urinary frequency >= 8 per day and urgency urinary incontinence >=1 per day

Exclusion Criteria:

* Patients with conditions that would contraindicate for fesoterodine use, e.g, hypersensitivity to the active substance (fesoterodine) or to peanut or soya or any of the excipients, urinary retention, and gastric retention.
* Patients with significant hepatic and renal disease or other significant unstable diseases.
* OAB symptoms caused by neurological conditions, known pathologies of urinary tract, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1712 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (156):
- United States (39):
  - Pfizer Investigational Site, Homewood, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Coeur d'Alene, Idaho
  - Pfizer Investigational Site, Sandpoint, Idaho
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, West Des Moines, Iowa
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Shrevport, Louisiana
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Lawrenceville, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Concord, North Carolina
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Menomonee Falls, Wisconsin
- Belgium (4):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Kortrijk
  - Pfizer Investigational Site, Tessenderlo
- Brazil (5):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Chile (3):
  - Pfizer Investigational Site, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Pfizer Investigational Site, Port Montt
  - Pfizer Investigational Site, Santiago
- Pfizer Investigational Site, Bogota, Cundinamarca, Colombia
- Costa Rica (3):
  - Pfizer Investigational Site, Alajuela, Alajuela Province
  - Pfizer Investigational Site, Cartago, Cartago Province
  - Pfizer Investigational Site, San José, Provincia de San José
- Czechia (5):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Jablonec nad Nisou
  - Pfizer Investigational Site, Jindřichův Hradec
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Prague
- Denmark (7):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Aarhus N
  - Pfizer Investigational Site, Glostrup Municipality
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Kolding
  - Pfizer Investigational Site, Nykoebing Falster
  - Pfizer Investigational Site, Roskilde
- Germany (10):
  - Pfizer Investigational Site, Ahaus
  - Pfizer Investigational Site, Alzey
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Krumbach
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Muelheim A.d. Ruhr
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Rosenheim
- Greece (4):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Ioannina, Ipiros
  - Pfizer Investigational Site, Rio, Patras
  - Pfizer Investigational Site, Thessaloniki
- Hong Kong (2):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Shatin
- Hungary (4):
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szentes
- India (5):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Vellore, Tamil Nadu
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Italy (3):
  - Pfizer Investigational Site, Latina
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Siena
- Malaysia (2):
  - Pfizer Investigational Site, Batu Caves, Selangor
  - Pfizer Investigational Site, Kuala Lumpur
- Norway (5):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Hamar
  - Pfizer Investigational Site, Lysaker
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Sandnes
- Peru (2):
  - Pfizer Investigational Site, Lima, Lima Province
  - Pfizer Investigational Site, Surco, Lima region
- Poland (5):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Romania (4):
  - Pfizer Investigational Site, Arad
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Sibiu
  - Pfizer Investigational Site, Timișoara
- Russia (4):
  - Pfizer Investigational Site, Moscow, Russia
  - Pfizer Investigational Site, Saint Petersburg, Russia
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- South Africa (7):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Parktown, Gauteng
  - Pfizer Investigational Site, Vosloorus, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Pietermaritzburg, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Pretoria
- South Korea (3):
  - Pfizer Investigational Site, Seoul, Korea
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Seoul
- Spain (4):
  - Pfizer Investigational Site, Getafe, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Bilbao, Vizcaya
- Sweden (5):
  - Pfizer Investigational Site, Huskvarna
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Switzerland (2):
  - Pfizer Investigational Site, Frauenfeld
  - Pfizer Investigational Site, Lucerne
- Taiwan (4):
  - Pfizer Investigational Site, Niao-Sung Hsiang, Kaohsiung
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Ukraine (5):
  - Pfizer Investigational Site, Chernivtsi
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Zaporizhzhia

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- [Derived] Corcos J, Angulo JC, Garely AD, Carlsson M, Gong J, Guan Z; Fesoterodine Assessment and Comparison Versus Tolterodine (FACT) Study Group. Effect of fesoterodine 4 mg on bladder diary and patient-reported outcomes during the first week of treatment in subjects with overactive bladder. Curr Med Res Opin. 2011 May;27(5):1059-65. doi: 10.1185/03007995.2011.565044. Epub 2011 Mar 23. PMID 21428726
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221008&StudyName=Clinical%20Trial%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Fesoterodine%20in%20Comparison%20to%20Tolterodine%20for%20Overactive%20Bladder

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with urgency incontinence Overactive Bladder (OAB) symptoms who met all entrance criteria were randomized to the double-blind treatment period.
Groups:
- Placebo: Tablets (4 milligrams [mg] orally (PO) once daily (QD) for 1 week followed by a forced dose escalation to 8 mg PO QD for 11 weeks) or capsules (4 mg) PO QD for 12 weeks
- Tolterodine ER: Capsules (4 mg) PO QD for 12 weeks. Tolterodine Extended Release (ER)
- Fesoterodine: Tablets (4 mg PO QD for 1 week followed by a forced dose escalation to 8 mg PO QD for 11 weeks)
Period: Single-blind Placebo Run-In Period
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Started | 2446 | 0 | 0
Completed | 1712 (progressed to randomization in double-blind treatment period) | 0 | 0
Not Completed | 734 | 0 | 0
Period: Randomized to Double-blind Treatment
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Started | 337 | 690 | 685
Completed | 334 | 684 | 679
Not Completed | 3 | 6 | 6
Not completed — Never returned after randomization | 3 | 6 | 6
Period: Double-blind Treatment Period
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Started | 334 | 684 | 679
Completed | 304 | 628 | 598
Not Completed | 30 | 56 | 81
Not completed — Death | 2 | 0 | 0
Not completed — Adverse Event | 6 | 28 | 44
Not completed — Lack of Efficacy | 5 | 5 | 13
Not completed — Lost to Follow-up | 4 | 8 | 5
Not completed — Withdrawal by Subject | 6 | 8 | 7
Not completed — Other | 7 | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tolterodine ER | Fesoterodine | Total
Number analyzed (Participants) | 334 | 684 | 679 | 1697
Age, Customized [Number; unit: participants]
  18 - 44 years | 55 | 103 | 96 | 254
  45 - 64 years | 167 | 349 | 367 | 883
  >= 65 years | 112 | 232 | 216 | 560
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 564 | 558 | 1391
  Male | 65 | 120 | 121 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12 (End of Treatment).
Description: UUI per 24 hours: total number of micturitions with Urinary Sensation Scale (USS) of 5 divided by total number of diary days collected at visit. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change: mean at observation minus mean at baseline.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS): took at least 1 dose of assigned treatment, contributed data to at least 1 baseline or post-baseline efficacy assessment, and excluded 107 subjects from two study sites with significant Good Clinical Practices (GCP) deviations. The decision to exclude that data was made while the study was still blinded.
Measure: Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 307 | 626 | 619
number of episodes per 24 hours | -1.46 (0.10) | -1.61 (0.06) | -1.72 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine versus (vs) placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the fifth (5th) and ninety-fifth (95th) percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test — Comparison fesoterodine vs tolterodine ER performed only if statistical significance favoring fesoterodine achieved for fesoterodine vs placebo to preserve overall alpha level at 5%; pairwise comparison also performed for tolterodine ER vs placebo; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0107, Van Elteren's Test — [p-value comment as in outcome 1, analysis 1]; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0172, Van Elteren's Test — [p-value comment as in outcome 1, analysis 1]; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile

2. Secondary Outcome: Change From Baseline in Mean Number of UUI Episodes Per 24 Hours at Week 1 and Week 4.
Description: UUI episodes per 24 hours calculated as total number of micturitions with Urinary Sensation Scale (USS) of 5 divided by total number of diary days collected at visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4
Population: FAS; Subjects reporting this symptom at baseline; (n)=number of subjects with baseline UUI>0 per 24 hours, non-missing change from baseline to respective post-baseline value (Week 1 or Week 4 [Last Observation Carried Forward (LOCF)]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
number of episodes per 24 hours
  Week 1 (n=302, 614, 612) | -0.54 (0.09) | -0.92 (0.06) | -0.95 (0.06)
  Week 4 [LOCF] (n=307, 626, 618) | -1.06 (0.10) | -1.40 (0.06) | -1.52 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.8460, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.1937, Van Elteren's Test; P-value based on Van Elteren's Test adjusted by baseline UUI quartile

3. Secondary Outcome: Percent Change From Baseline of UUI Episodes Per 24 Hours.
Description: UUI episodes per 24 hours calculated as total number of micturitions with USS of 5 in diary. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as UUI episodes per 24 hours at observation divided by baseline number of UUI episodes per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; Subjects reporting this symptom at baseline; (n)=number of subjects with baseline UUI>0 per 24 hours, non-missing change from baseline to respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
percent change
  Week 1 (n=302, 614, 612) | -28.6 [-100.0 to 300.0] | -55.1 [-100.0 to 537.5] | -53.6 [-100.0 to 525.0]
  Week 4 [LOCF] (n=307, 626, 618) | -60.0 [-100.0 to 300.0] | -85.7 [-100.0 to 650.0] | -93.2 [-100.0 to 450.0]
  Week 12 [LOCF] (n=307, 626, 619) | -82.1 [-100.0 to 300.0] | -100.0 [-100.0 to 450.0] | -100.0 [-100.0 to 400.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 1: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — Inferential testing: percent change from baseline only carried out for given end/time point if corresponding numeric change result statistically significant (to preserve alpha level at 5% within each type of diary endpoint for a given comparison); Based on a ranked analysis of covariance model with country and treatment as factors, and ranked baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 1: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 4: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 4: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0220, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition.
Description: Mean voided volume calculated as sum of voided volume divided by the total number of micturition episodes with a recorded voided volume greater than 0 in the 3-day diary at that visit.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of subjects with non-missing numerical change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: voided volume per micturition
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
voided volume per micturition
  Week 1 (n=306, 622, 623) | 11.0 (3.2) [5.0 to 14.5] | 19.2 (2.5) [13.6 to 21.3] | 18.7 (2.5) [12.6 to 20.9]
  Week 4 [LOCF] (n=313, 633, 625) | 14.0 (3.8) [6.9 to 18.9] | 25.7 (3.0) [19.4 to 29.0] | 30.5 (3.0) [24.0 to 33.3]
  Week 12 [LOCF] (n=313, 633, 626) | 16.8 (3.9) [9.9 to 22.7] | 23.5 (3.0) [17.1 to 26.9] | 32.9 (3.1) [26.1 to 35.8]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0214, ANCOVA; Based on an analysis of covariance model with country and treatment as factors, and centered baseline value as a covariate; Mean Difference (Final Values) = 7.8, Standard Error of Mean 3.4 — Treatment Difference Least Squares Mean (LSMean) Difference Standard Error (SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0149, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 8.2, Standard Error of Mean 3.4 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.8659, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.5, Standard Error of Mean 2.7 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 16.5, Standard Error of Mean 4.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0036, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 11.7, Standard Error of Mean 4.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.1484, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 4.7, Standard Error of Mean 3.3 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 16.1, Standard Error of Mean 4.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.1029, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 6.7, Standard Error of Mean 4.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0048, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 9.4, Standard Error of Mean 3.3 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

5. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours.
Description: The mean number of micturitions was calculated as the sum of all micturitions divided by the total number of diary days collected at that visit. Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: number of micturitions per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
number of micturitions per 24 hours
  Week 1 (n=307, 622, 623) | -0.5 (0.1) | -1.0 (0.1) | -1.0 (0.1)
  Week 4 [LOCF] (n= 313, 634, 627) | -1.2 (0.2) | -1.8 (0.1) | -1.9 (0.1)
  Week 12 [LOCF] (n= 313, 634, 628) | -1.5 (0.2) | -2.1 (0.1) | -2.2 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.5, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.7395, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.0, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0007, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.4185, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0005, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.3798, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

6. Secondary Outcome: Percent Change From Baseline of Micturitions Per 24 Hours.
Description: Percent change of micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (ie, 100% *(Week 12 or 4 - baseline)/baseline).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of subjects with non-missing percent change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
percent change
  Week 1 (n=307, 622, 623) | -2.7 [-48.5 to 68.3] | -7.7 [-68.2 to 70.0] | -7.9 [-66.0 to 184.0]
  Week 4 [LOCF] (n=313, 634, 627) | -10.3 [-67.4 to 75.0] | -15.0 [-66.2 to 82.9] | -14.8 [-67.6 to 135.7]
  Week 12 [LOCF] (n=313, 634, 628) | -12.1 [-69.6 to 73.0] | -16.2 [-69.6 to 55.6] | -18.9 [-66.7 to 185.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 12: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12. Per closed testing procedure, statistical testing for percent change not performed for Fesoterodine vs Tolterodine ER Week 12: corresponding numerical change result not statistically significant; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturitions Per 24 Hours.
Description: Mean number of nocturnal micturitions per 24 hours was calculated as the sum of all micturitions divided by the total number of diary days collected at that visit. Nocturnal (Bedtime) was defined as the time the subject went to bed until he/she arose to start the next day.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; Subjects reporting this symptom at baseline; (n)=number of subjects with baseline nocturnal micturitions >0 per 24 hours, non-missing change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: nocturnal micturitions per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
nocturnal micturitions per 24 hours
  Week 1 (n=288, 584, 596) | -0.1 (0.1) | -0.3 (0.0) | -0.2 (0.0)
  Week 4 [LOCF] (n=293, 596, 600) | -0.4 (0.1) | -0.5 (0.0) | -0.5 (0.1)
  Week 12 [LOCF] (n=293, 596, 601) | -0.5 (0.1) | -0.6 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.2730, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0652, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.3503, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.0, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p = 0.2667, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.1643, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.7264, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.0, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.3269, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.5059, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.0, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.6990, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.0, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

8. Secondary Outcome: Percent Change From Baseline of Nocturnal Micturitions Per 24 Hours.
Description: Percent change of nocturnal micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (ie, 100% *(Week 12 or 4 - baseline)/baseline). Nocturnal (Bedtime) was defined as the time the subject went to bed until he/she arose to start the next day.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
percent change
  Week 1 (n=288, 584, 596) | -10.0 [-100.0 to 500.0] | -12.5 [-100.0 to 350.0] | 0.0 [-100.0 to 800.0]
  Week 4 [LOCF] (n=293, 596, 600) | -22.2 [-100.0 to 600.0] | -25.0 [-100.0 to 400.0] | -20.0 [-100.0 to 900.0]
  Week 12 [LOCF] (n=293, 596, 601) | -25.0 [-100.0 to 600.0] | -27.9 [-100.0 to 500.0] | -28.6 [-100.0 to 400.0]

9. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours.
Description: Mean number urgency episodes (USS rating >= to 3 in diary) per 24 hours calculated as sum of all micturitions divided by total number of diary days collected at visit. USS: 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; Subjects reporting this symptom at baseline; (n)=number of subjects with baseline urgency episodes >0 per 24 hours, non-missing change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
urgency episodes per 24 hours
  Week 1 (n=306, 619, 621) | -0.4 (0.2) | -1.3 (0.2) | -1.1 (0.2)
  Week 4 [LOCF] (n=311, 631, 627) | -1.2 (0.2) | -2.4 (0.2) | -2.6 (0.2)
  Week 12 [LOCF] (n=311, 631, 628) | -2.0 (0.3) | -3.1 (0.2) | -3.5 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0008, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.3820, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.4, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.2, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.3498, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.5, Standard Error of Mean 0.3 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.1, Standard Error of Mean 0.3 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0542, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.4, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

10. Secondary Outcome: Percent Change From Baseline of Urgency Episodes Per 24 Hours.
Description: Percent change of urgency episodes (USS rating >= to 3 in diary) per 24 hours calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100. USS: 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 9
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
percent change
  Week 1 (n=306, 619, 621) | -5.6 [-100.0 to 271.4] | -12.5 [-100.0 to 400.0] | -9.7 [-100.0 to 485.7]
  Week 4 [LOCF] (n=311,631, 627) | -11.4 [-100.0 to 560.0] | -23.1 [-100.0 to 233.3] | -26.9 [-100.0 to 385.7]
  Week 12 [LOCF] (n=311, 631, 628) | -17.6 [-100.0 to 560.0] | -30.8 [-100.0 to 372.7] | -37.9 [-100.0 to 385.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

11. Secondary Outcome: Change From Baseline in Mean Number of Severe Urgency Episodes Per 24 Hours.
Description: Mean number of severe urgency episodes (USS rating >= to 4 in diary ) per 24 hours: sum of all micturitions divided by total number of diary days collected at that visit. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; Subjects reporting this symptom at baseline; (n)=number of subjects with baseline severe urgency episodes >0 per 24 hours, non-missing change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: severe urgency episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
severe urgency episodes per 24 hours
  Week 1 (n=306, 618, 618) | -0.4 (0.2) | -1.3 (0.2) | -1.2 (0.2)
  Week 4 [LOCF] (n=311, 630, 624) | -1.2 (0.2) | -2.2 (0.2) | -2.4 (0.2)
  Week 12 [LOCF] (n=311, 630, 625) | -1.9 (0.2) | -2.8 (0.2) | -3.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.0, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.5581, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.1, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.2, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.0, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.1510, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.1, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.1391, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

12. Secondary Outcome: Percent Change From Baseline of Severe Urgency Episodes Per 24 Hours.
Description: Percent change calculated as change in severe urgency episodes (USS rating >= to 4 in diary ) per 24 hours at that visit divided by the baseline number of severe urgency episodes per 24 hours, multiplied by 100. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 11
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
percent change
  Week 1 (n=306, 618, 618) | -9.4 [-100.0 to 500.0] | -25.0 [-100.0 to 775.0] | -25.0 [-100.0 to 680.0]
  Week 4 [LOCF] (n=311, 630, 624) | -25.0 [-100.0 to 866.7] | -45.8 [-100.0 to 460.0] | -54.5 [-100.0 to 550.0]
  Week 12 [LOCF] (n=311, 630, 625) | -48.0 [-100.0 to 733.3] | -63.4 [-100.0 to 412.5] | -71.4 [-100.0 to 585.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

13. Secondary Outcome: Change From Baseline in Mean USS Rating Per Micturition Per 24 Hours.
Description: Mean USS rating calculated as the sum of rating scores on USS per 24 hours divided by the mean number of micturitions per 24 hours at that visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
score on scale
  Week 1 (n=306, 619, 621) | -0.1 (0.0) | -0.2 (0.0) | -0.2 (0.0)
  Week 4 [LOCF] (n=311, 631, 627) | -0.2 (0.0) | -0.4 (0.0) | -0.5 (0.0)
  Week 12 [LOCF] (n=311, 631, 628) | -0.4 (0.0) | -0.6 (0.0) | -0.7 (0.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.5972, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.0, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.1267, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.1 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0289, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.0 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

14. Secondary Outcome: Change From Baseline in Frequency-Urgency Sum (Formerly Known as Urinary Sensations Scale Sum in Protocol) Per 24 Hours.
Description: Frequency-Urgency Sum rating per 24 hours calculated as mean rating scores on the USS multiplied by the mean number of micturitions per 24 hours at that visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as mean at observation minus mean at baseline.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
score on scale
  Week 1 (n=306, 619, 621) | -2.4 (0.7) | -5.7 (0.5) | -5.5 (0.5)
  Week 4 [LOCF] (n=311,631, 627) | -5.7 (0.8) | -9.7 (0.6) | -10.5 (0.6)
  Week 12 [LOCF] (n=311, 631, 628) | -8.2 (0.8) | -12.1 (0.6) | -13.2 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.1, Standard Error of Mean 0.7 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.3, Standard Error of Mean 0.7 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.7288, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.6 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -4.7, Standard Error of Mean 0.8 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -4.0, Standard Error of Mean 0.8 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.2473, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.6 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -4.9, Standard Error of Mean 0.8 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.8, Standard Error of Mean 0.8 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.1047, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.1, Standard Error of Mean 0.7 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

15. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC).
Description: Number of subjects in 4-point category: >= to 2 points improvement [major improvement]; 1 point improvement [minor improvement]; no change; deterioration, based on PPBC score (rated on 6-point scale: 1=no problems at all; 6=many severe problems). Score change: score at observation minus score at baseline; re-scaled to 4-point categorical variables.
Time Frame: Baseline, Week 1, Week, 4, Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
participants
  Week 1 (n=309, 625, 623), >=2 points improvement | 32 | 79 | 102
  Week 1, 1-point improvement | 94 | 181 | 186
  Week 1, no change | 147 | 306 | 286
  Week 1, deterioration | 36 | 59 | 49
  Week 4 (n=313, 632, 629), >=2 points improvement | 57 | 169 | 196
  Week 4, 1-point improvement | 95 | 201 | 224
  Week 4, no change | 127 | 203 | 176
  Week 4, deterioration | 34 | 59 | 33
  Week 12 (n=313, 632, 630), >=2 points improvement | 67 | 210 | 254
  Week 12, 1-point improvement | 102 | 189 | 198
  Week 12, no change | 111 | 171 | 148
  Week 12, deterioration | 33 | 62 | 30
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0143, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country

16. Secondary Outcome: Change From Baseline in Urgency Perception Scale (UPS). UPS Equals Patient Perception of Urgency Scale (PPUS) in Protocol.
Description: Number of subjects in 3-point category: improvement [>=1-point improvement]; no change; deterioration [>=1-point decrease], based on UPS score (rated on 3-point scale: 1=not able to hold urine; 3=able to finish what I am doing). Score change calculated as score at observation minus score at baseline; re-scaled to 3-point categorical variables.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
participants
  Week 1 (n=309, 627, 624), improvement | 68 | 162 | 171
  Week 1, no change | 218 | 438 | 413
  Week 1, deterioration | 23 | 27 | 40
  Week 4 (n=313, 633, 629), improvement | 98 | 238 | 256
  Week 4, no change | 194 | 362 | 348
  Week 4, deterioration | 21 | 33 | 25
  Week 12 (n=313, 633, 630), improvement | 112 | 254 | 291
  Week 12, no change | 181 | 344 | 314
  Week 12, deterioration | 20 | 35 | 25
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0773, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; With modified ridit scoring and stratified by country

17. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q): Symptom Bother Score at Week 12 (End of Treatment).
Description: Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/by raw score range * 100]. Higher transformed scores indicative of greater symptom bother. Negative change in Symptom Bother score indicates improvement. Change calculated as score at observation minus score at baseline.
Time Frame: Baseline, Week 12
Population: FAS; (n)=number of subjects with non-missing numerical change from baseline to Week 12 for placebo n=289; Tolterodine ER n=589; Fesoterodine n=571.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
score on scale | -16.3 (1.4) | -22.5 (1.1) | -27.1 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -10.8, Standard Error of Mean 1.5 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

18. Secondary Outcome: Change From Baseline in OAB-q: Health Related Quality of Life (HRQL) at Week 12 (End of Treatment).
Description: HRQL domain and total raw score derived as sum of scores (6-point scale: 1=not at all/none of the time; 6=a very great deal/all of the time). Transformed score (Total HRQL or domain)=[(Highest possible raw score-Actual total raw score)/Raw score range]x100. Higher transformed scores indicative of better HRQL. Positive change in HRQL scores indicates improvement. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 12
Population: FAS; (n)=number of subjects with non-missing numerical change from baseline to Week 12 for placebo, Tolterodine ER, and Fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
score on scale
  HRQL concern domain (n=289, 589, 572) | 13.4 (1.5) | 19.3 (1.1) | 22.6 (1.2)
  HRQL coping domain (n=289, 589, 572) | 14.0 (1.5) | 18.5 (1.2) | 22.6 (1.2)
  HRQL sleep domain (n=289, 589, 572) | 12.2 (1.4) | 15.1 (1.1) | 17.3 (1.1)
  HRQL social interaction domain (n=289, 588, 572) | 6.8 (1.1) | 9.4 (0.9) | 11.6 (0.9)
  HRQL scale score total (n=289, 588, 572) | 12.0 (1.3) | 16.3 (1.0) | 19.3 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL concern domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 9.2, Standard Error of Mean 1.6 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL coping domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 8.6, Standard Error of Mean 1.6 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL sleep domain; Test type: Superiority or Other; p = 0.0008, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 5.0, Standard Deviation 1.5 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL social interaction domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 4.8, Standard Error of Mean 1.2 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL scale score total; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 7.3, Standard Error of Mean 1.3 — Treatment Difference LSMean Difference(SE), SE is recorded as Parameter Dispersion Type: Standard Error of the mean

19. Post Hoc Outcome: Diary Dry Rates
Description: Diary dry rate: number of subjects with no urgency urinary incontinence episode reported in the 3 day diary at the respective time-point; based on USS: 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Week 1, Week 4, Week 12
Population: FAS; only subjects with baseline urgency urinary incontinence >0 per 24 hours are included; n=number of subjects in the respective category at observation (Week 1, Week 4, Week 12).
Measure: Number; unit: participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 334 | 684 | 679
participants
  Week 1 | 54 | 153 | 159
  Week 4 | 97 | 290 | 306
  Week 12 | 138 | 358 | 396
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0072, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0116, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.7828, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.3104, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0153, Cochran-Mantel-Haenszel; Stratified by baseline urgency urinary incontinence quartile

ADVERSE EVENTS:
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 8 | 9 | 15
Other Adverse Events (participants affected / at risk) | 76 | 213 | 290
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Tolterodine ER | Fesoterodine
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0/334 | 0/684 | 1/679
Hypertensive heart disease (Cardiac disorders) | 0/334 | 0/684 | 1/679
Myocardial ischaemia (Cardiac disorders) | 0/334 | 0/684 | 1/679
Abdominal pain (Gastrointestinal disorders) | 0/334 | 0/684 | 1/679
Appendicitis perforated (Gastrointestinal disorders) | 0/334 | 0/684 | 1/679
Nausea (Gastrointestinal disorders) | 1/334 | 0/684 | 0/679
Rectal haemorrhage (Gastrointestinal disorders) | 0/334 | 0/684 | 1/679
Vomiting (Gastrointestinal disorders) | 1/334 | 0/684 | 0/679
Chest pain (General disorders) | 0/334 | 1/684 | 0/679
Biliary colic (Hepatobiliary disorders) | 0/334 | 1/684 | 0/679
Abdominal wall abscess (Infections and infestations) | 1/334 | 0/684 | 0/679
Bronchiectasis (Infections and infestations) | 0/334 | 0/684 | 1/679
Cystitis (Infections and infestations) | 0/334 | 1/684 | 0/679
Herpes zoster (Infections and infestations) | 0/334 | 1/684 | 0/679
Hand fracture (Injury, poisoning and procedural complications) | 1/334 | 0/684 | 0/679
Head injury (Injury, poisoning and procedural complications) | 0/334 | 1/684 | 0/679
Seroma (Injury, poisoning and procedural complications) | 1/334 | 0/684 | 0/679
Traumatic brain injury (Injury, poisoning and procedural complications) | 0/334 | 0/684 | 1/679
Upper limb fracture (Injury, poisoning and procedural complications) | 0/334 | 0/684 | 1/679
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/334 | 0/684 | 0/679
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/334 | 1/684 | 1/679
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/334 | 0/684 | 0/679
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/334 | 0/684 | 0/679
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/334 | 0/684 | 0/679
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/334 | 1/684 | 0/679
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/334 | 0/684 | 1/679
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/334 | 0/684 | 0/679
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/334 | 1/684 | 0/679
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/334 | 0/684 | 0/679
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/334 | 0/684 | 1/679
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/334 | 0/684 | 0/679
Dizziness (Nervous system disorders) | 1/334 | 0/684 | 0/679
Haemorrhage intracranial (Nervous system disorders) | 0/334 | 0/684 | 1/679
Vertebrobasilar insufficiency (Nervous system disorders) | 1/334 | 0/684 | 0/679
Mental status changes (Psychiatric disorders) | 1/334 | 0/684 | 0/679
Suicidal behaviour (Psychiatric disorders) | 0/334 | 0/684 | 1/679
Urinary incontinence (Renal and urinary disorders) | 0/334 | 0/684 | 1/679
Breast mass (Reproductive system and breast disorders) | 0/334 | 1/684 | 0/679
Uterine haemorrhage (Reproductive system and breast disorders) | 0/334 | 0/684 | 1/679
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/334 | 0/684 | 0/679
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/334 | 1/684 | 0/679
Arteriosclerosis (Vascular disorders) | 1/334 | 0/684 | 0/679
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Tolterodine ER | Fesoterodine
Dry eye (Eye disorders) | 6/334 | 8/684 | 9/679
Vision blurred (Eye disorders) | 1/334 | 8/684 | 12/679
Abdominal pain (Gastrointestinal disorders) | 4/334 | 4/684 | 10/679
Abdominal pain upper (Gastrointestinal disorders) | 3/334 | 6/684 | 9/679
Constipation (Gastrointestinal disorders) | 10/334 | 28/684 | 37/679
Diarrhoea (Gastrointestinal disorders) | 4/334 | 15/684 | 14/679
Dry mouth (Gastrointestinal disorders) | 20/334 | 112/684 | 189/679
Dyspepsia (Gastrointestinal disorders) | 1/334 | 8/684 | 12/679
Nausea (Gastrointestinal disorders) | 6/334 | 7/684 | 12/679
Vomiting (Gastrointestinal disorders) | 2/334 | 2/684 | 7/679
Fatigue (General disorders) | 0/334 | 4/684 | 12/679
Influenza (Infections and infestations) | 4/334 | 8/684 | 7/679
Nasopharyngitis (Infections and infestations) | 10/334 | 13/684 | 13/679
Sinusitis (Infections and infestations) | 3/334 | 8/684 | 3/679
Upper respiratory tract infection (Infections and infestations) | 4/334 | 9/684 | 2/679
Urinary tract infection (Infections and infestations) | 2/334 | 10/684 | 15/679
Back pain (Musculoskeletal and connective tissue disorders) | 10/334 | 7/684 | 10/679
Dizziness (Nervous system disorders) | 3/334 | 10/684 | 8/679
Headache (Nervous system disorders) | 8/334 | 23/684 | 38/679
Dysuria (Renal and urinary disorders) | 1/334 | 7/684 | 4/679
Cough (Respiratory, thoracic and mediastinal disorders) | 1/334 | 4/684 | 8/679
Hypertension (Vascular disorders) | 3/334 | 3/684 | 8/679

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.